CLINICAL TRIAL: NCT01910194
Title: A Bicentric Open-label, Randomized, Two-parallel-group Study Investigating the Impact of Combined Lantus Insulin Glargine) and Lyxumia(Lixisenatide) on Insulin Secretion and Gastric Emptying in Subjects With Type 2 Diabetes Mellitus Not Adequately Controlled on Diet and Oral Antidiabetic Medication
Brief Title: Impact of Combined of Lantus(Insulin Glargine) and Lyxumia (Lixisenatide) on Insulin Secretion and Gastric Emptying
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: LanLyx
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lyxumia (Other): 4 weeks Luxumia plus another 4 weeks combination
  Interventions: Drug: Luyxumia versus Lantus
- Lantus (Other): 4 weeks Lantus plus another 4 weeks combination
  Interventions: Drug: Luyxumia versus Lantus

INTERVENTIONS:
Drug: Luyxumia versus Lantus

SUMMARY:
Impact of combined Lantus (insulin glargine) and Lyxumia(lixisenatide) on insulin secretion and gastric emptying

DETAILED DESCRIPTION:
Impact of combined Lantus (insulin glargine) and Lyxumia(lixisenatide) on insulin secretion and gastric emptying

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus diagnosed at least one year before the screening visit not previously treated with glitazones, insulin or GLP-1 agonists
* Inadequately controlled diabetes mellitus

Exclusion Criteria:

* Subjects with type 1 diabetes, maturity onset diabetes of the young (MODY) or secondary forms of diabetes such as due to pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
AUCISEC(0-10min) | Within 0 to 10 min after iv glucose challenge

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - St. Josef-Hospital, University Hospital, Ruhr, Bochum
  - Profil Institut für Stoffwechselforschung GmbH, Neuss